CLINICAL TRIAL: NCT00088205
Title: A Phase 2 Study of Oral Enzastaurin HCl in Patients With Relapsed Mantle Cell Lymphoma
Brief Title: Oral Enzastaurin in Participants With Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8360; H6Q-MC-JCAO (Other: Eli Lilly and Company)
Record Dates: First submitted 2004-07-22; First posted 2004-07-23 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Mantle-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: enzastaurin

INTERVENTIONS:
Drug: enzastaurin — 500 milligrams (mg), oral, daily, up to six 28-day cycles
  Other Names: LY317615

SUMMARY:
The purposes of this study are to determine the safety of oral enzastaurin and any side effects that might be associated with it and whether enzastaurin can help participants with mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Mantle cell lymphoma
* Previous treatment for mantle cell lymphoma
* Previously relapsed mantle cell lymphoma with no more than 4 chemotherapy regimens.
* Have discontinued all previous therapies for cancer, except corticosteroids up to 25 milligrams per day (mg/day)
* Adequate organ function

Exclusion Criteria:

* Inability to swallow tablets
* Must not have significant heart problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Woolloongabba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Parkville, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Prahran, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Wodonga, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, East Melbourne
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rouen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tours
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Homburg Saar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kassel
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rotterdam

REFERENCES:
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reports those participants who discontinued from study drug. Only participants without confirmed progressive disease at the 30-day post-therapy visit were assessed for progression by radiological method every 3 months until disease progression.
Groups:
- Enzastaurin: 500 milligrams (mg) oral dose administered once daily, in the morning, during each 28-day cycle of therapy for planned duration of treatment up to 6 cycles in the absence of disease progression or for any other cause of discontinuation. Treatment was continued until unacceptable toxicity or progressive disease occurred.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 60
Received at Least 1 Dose of Study Drug | 60
Efficacy Population | 59 (Participants with diagnosis of relapsed mantle cell lymphoma.)
Completed | 0
Not Completed | 60
Not completed — Adverse Event | 4
Not completed — Progressive Disease | 51
Not completed — Physician Decision | 1
Not completed — Death Due to Study Disease | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Enzastaurin: 500 mg oral dose administered once daily, in the morning, during each 28-day cycle of therapy for planned duration of treatment up to 6 cycles in the absence of disease progression or for any other cause of discontinuation. Treatment was continued until unacceptable toxicity or progressive disease occurred.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 66.0 [45.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  France | 28
  Australia | 12
  Germany | 13
  Netherlands | 7
Baseline B Symptoms [Count of Participants; unit: Participants] — B symptoms include weight loss >10% of body weight in the preceding 6 months, unexplained fevers >38°C, drenching night sweats and assigned an international prognostic index score of low (0-1), medium (2-3) or high (4-5). Higher scores indicate worse symptoms.
  Participants
    Low (0-1) | 9
    Medium (2-3) | 39
    High (4-5) | 8
    Not available | 4
Participants with High Lactate Dehydrogenase (LDH) [Count of Participants; unit: Participants] — Participants with LDH >300 international units/liter (IU/L) are considered having high LDH.
  Participants | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Progression (FFP) for at Least 3 Cycles
Description: Using the Standardized Response Criteria for non-Hodgkin's lymphomas, participants were considered to have progressive disease if there was a 50% increase in the sum of the products of the greatest diameters (SPD) of the dominant nodal and non-nodal sites or appearance of new-involved site or lesion. The percentage of FFP was computed as the number of participants documented to be progression free after 3 cycles of treatment divided by the number of treated participants and then multiplied by 100.
Time Frame: Baseline through at least 3 cycles of treatment (28-day cycle)
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 59
percentage of participants | 35.6 [23.4 to 47.8]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) Plus Unconfirmed Complete Response (CRu) Plus Partial Response (PR) (Objective Response Rate)
Time Frame: Baseline to 22.01 months
Population: Zero participants were analyzed as no participant achieved CR, CRu or PR.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS time was defined as the time from the date of enrollment to the first date of documented progressive disease or death due to any cause, whichever occurred first. Using the Standardized Response Criteria for non-Hodgkin's lymphomas, participants were considered to have progressive disease if there was a 50% increase in the sum of the products of the greatest diameters (SPD) of the dominant nodal and non-nodal sites or appearance of new-involved site or lesion. Progression-free survival time was censored at the date of the last assessment visit for participants who were still alive and who had not had documented progressive disease.
Time Frame: Baseline to measured progressive disease or death due to any cause up to 22.01 months
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug. Participants censored = 3.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 59
months | 1.97 [1.45 to 2.66]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of enrollment to the date of death due to any cause. For each participant who was not known to have died as of the data-inclusion cut-off date, OS was censored for that analysis at the date of the last assessment visit prior to the cut-off date.
Time Frame: Baseline to date of death from any cause at least up to 23.10 months
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug. Participants censored = 39.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 59
months | 22.01 [13.93 to NA] — Upper limit of 95% Confidence Interval was not estimable due to high censoring rate.

5. Secondary Outcome: Duration of CR, CRu, PR or Stable Disease (SD) [Duration of Overall Response]
Description: Duration of overall response for responders was measured from the date that measurement criteria were met for CR, CRu, PR or SD (whichever status occurred first) until the first date of documented progressive disease or death due to any cause, whichever occurred first. Using the Standardized Response Criteria for non-Hodgkin's lymphomas Guidelines, CR was defined as the disappearance of all lesions. CRu was the disappearance of clinical and radiographic evidence of disease, normal appearance of spleen and greater than 75% regression in lymph node mass. PR was defined as at least a 50% decrease in the six largest dominant nodes. SD was when the response was poorer than partial response with no new lesions consistent with progressive disease. Duration of response was censored at the date of the last assessment visit for responders who were still alive and had not had documented progressive disease.
Time Frame: Date of progression or death due to any cause up to 22.01 months
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug and met criteria for CR, CRu, PR or SD. Participants censored = 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 13
months | 5.55 [4.67 to 8.15]

6. Secondary Outcome: Time to New Treatment
Description: Time to new treatment was as the time from enrollment to the date new treatment for the cancer under study was initiated. Time to new treatment was censored at the date of the last assessment visit for participants who were not documented to have initiated a new treatment.
Time Frame: Baseline to date of new treatment up to 23.10 months
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug. Participants censored =16.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 59
months | 3.52 [2.37 to 4.04]

7. Secondary Outcome: Change in Scores From Baseline to Cycle 6 in Functional Assessment of Cancer Therapy Lymphoma Version 4 ( FACT-Lym v.4)
Description: The B symptoms, tumor-related symptoms, participant functioning, and health-related quality of life were assessed with FACT-Lym v. 4. FACT-Lym v. 4 consists of 42 items with 5-point rating scales for each item, where 0 = "not at all" and 4 = "very much." Physical well-being, social/family well-being and functional well-being subscales consist of 7 items each with scores ranging from 0-28. The emotional well-being subscale consists of 6 items with a score ranging from 0-24. The lymphoma tumor - specific subscale consists of 15 items with a score ranging from 0-60. Fact-Lymphoma total score ranges from 0-168. A higher score represents better quality of life.
Time Frame: Baseline, Cycles 2, 4 and 6 (28-day cycle)
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug and had FACT-Lym assessed at baseline and Cycles 2, 4 and 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin
Number analyzed (Participants) | 59
units on a scale
  Physical Well-being- Baseline: number analyzed (Participants) | 58
  Physical Well-being- Baseline | 22.45 (4.298)
  Physical Well-being- Cycle 2: number analyzed (Participants) | 39
  Physical Well-being- Cycle 2 | 22.06 (4.49)
  Physical Well-being- Cycle 4: number analyzed (Participants) | 18
  Physical Well-being- Cycle 4 | 22.15 (4.52)
  Physical Well-being- Cycle 6: number analyzed (Participants) | 10
  Physical Well-being- Cycle 6 | 21.6 (3.406)
  Social Family Well-being- Baseline: number analyzed (Participants) | 58
  Social Family Well-being- Baseline | 21.13 (4.792)
  Social Family Well-being- Cycle 2: number analyzed (Participants) | 39
  Social Family Well-being- Cycle 2 | 20.32 (6.165)
  Social Family Well-being- Cycle 4: number analyzed (Participants) | 18
  Social Family Well-being- Cycle 4 | 19.2 (5.421)
  Social Family Well-being- Cycle 6: number analyzed (Participants) | 10
  Social Family Well-being- Cycle 6 | 21.26 (4.021)
  Emotional Well-being- Baseline: number analyzed (Participants) | 58
  Emotional Well-being- Baseline | 17.41 (4.547)
  Emotional Well-being- Cycle 2: number analyzed (Participants) | 39
  Emotional Well-being- Cycle 2 | 17.65 (4.953)
  Emotional Well-being- Cycle 4: number analyzed (Participants) | 18
  Emotional Well-being- Cycle 4 | 17.56 (4.961)
  Emotional Well-being- Cycle 6: number analyzed (Participants) | 10
  Emotional Well-being- Cycle 6 | 17.25 (5.514)
  Functional Well-being- Baseline: number analyzed (Participants) | 58
  Functional Well-being- Baseline | 16.38 (5.768)
  Functional Well-being- Cycle 2: number analyzed (Participants) | 39
  Functional Well-being- Cycle 2 | 16.56 (6.05)
  Functional Well-being- Cycle 4: number analyzed (Participants) | 18
  Functional Well-being- Cycle 4 | 16.17 (4.076)
  Functional Well-being- Cycle 6: number analyzed (Participants) | 10
  Functional Well-being- Cycle 6 | 17.43 (4.871)
  Lymphoma Subscale- Baseline: number analyzed (Participants) | 58
  Lymphoma Subscale- Baseline | 46.27 (8.78)
  Lymphoma Subscale- Cycle 2: number analyzed (Participants) | 39
  Lymphoma Subscale- Cycle 2 | 46.01 (8.841)
  Lymphoma Subscale- Cycle 4: number analyzed (Participants) | 18
  Lymphoma Subscale- Cycle 4 | 46.9 (7.555)
  Lymphoma Subscale- Cycle 6: number analyzed (Participants) | 10
  Lymphoma Subscale- Cycle 6 | 46.8 (8.108)
  Fact-Lymphoma Total Score- Baseline: number analyzed (Participants) | 58
  Fact-Lymphoma Total Score- Baseline | 123.6 (22.21)
  Fact-Lymphoma Total Score- Cycle 2: number analyzed (Participants) | 39
  Fact-Lymphoma Total Score- Cycle 2 | 122.6 (23.8)
  Fact-Lymphoma Total Score- Cycle 4: number analyzed (Participants) | 18
  Fact-Lymphoma Total Score- Cycle 4 | 122 (20.67)
  Fact-Lymphoma Total Score- Cycle 6: number analyzed (Participants) | 10
  Fact-Lymphoma Total Score- Cycle 6 | 124.3 (21.92)

8. Secondary Outcome: Change From Baseline to Cycle 6 in European Quality of Life-5D (EuroQol-5D) Index Score (Overall Health Status)
Description: Overall health status and participant utility values were measured with the EuroQol-5D questionnaire. EuroQol-5D describes health status in terms of 5 dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension is divided into 3 levels: 1 (no problem), 2 (some problem), and 3 (extreme problem). The questionnaire records the level of problems on each of 5 dimensions and is converted into the EuroQol-5D index based on preference weights (Dolan 1997), where a score of 0.0 = death and 1.0 = perfect health.
Time Frame: Baseline, Cycles 2, 4 and 6
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug and had EuroQol-5D assessed at baseline and Cycles 2, 4, and 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin
Number analyzed (Participants) | 59
units on a scale
  Baseline: number analyzed (Participants) | 58
  Baseline | 0.70 (0.28)
  Cycle 2: number analyzed (Participants) | 36
  Cycle 2 | 0.76 (0.19)
  Cycle 4: number analyzed (Participants) | 18
  Cycle 4 | 0.74 (0.16)
  Cycle 6: number analyzed (Participants) | 10
  Cycle 6 | 0.68 (0.27)

9. Secondary Outcome: Number of Participants With Protein Kinase C Beta (PKCβ) Expression by Immunohistochemistry (IHC) Staining
Description: IHC staining of tumor samples was carried out to determine PKCβ expression. Staining intensity was measured on a semiquantitative scale of 0 (or negative) to 3 (high intensity). The final score combined the components of staining intensity and the percentage of positive cells and was defined as [1 * (percentage of cells staining at 1)] + [2 * (percentage of cells staining at 2)] + [3 * (percentage of cells staining at 3)]. Score ≥100 and staining intensity ≥2 indicates high expression for PKCβ, while score <100 and staining intensity ≤1 indicates low expression for PKCβ.
Time Frame: Baseline
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug and provided tissue specimens from the initial diagnosis for PKCβ expression analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 18
Participants
  Score ≥100 and staining intensity ≥2 | 14
  Score <100 and staining intensity ≤1 | 4

10. Secondary Outcome: Number of Participants With High Ki-67 Expression by IHC Staining
Description: IHC staining of tumor samples was carried out to determine Ki-67 expression. High expression is defined as the percentage of positive cells ≥40%.
Time Frame: Baseline
Population: All enrolled participants with relapsed mantle cell lymphoma who received at least 1 dose of study drug and provided tissue specimens from the initial diagnosis for Ki-67 expression analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
Participants | 4

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) (Safety of Enzastaurin)
Description: Data presented are the number of participants who experienced SAEs, AEs, deaths due to progressive disease (PD), and deaths due to AEs while on treatment and death during the 30-day post-treatment follow-up. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Each cycle (28-day cycle) up to 21 cycles and 30-day follow-up
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 60
Participants
  SAEs | 20
  Other non-serious AEs | 54
  Deaths due to PD | 4
  Deaths due to AEs | 0
  Deaths during 30-day follow-up | 6

12. Secondary Outcome: Average Steady-State Plasma Concentration (Cav,ss,) of Enzastaurin and Total Analytes (Pharmacokinetics of Enzastaurin and Total Analytes)
Description: The Steady-state plasma concentrations of total analytes (enzastaurin plus its active metabolite, LSN326020) observed after once-daily dosing were evaluated using sparse sampling methodology.
Time Frame: Cycles 1 [1-4 hours (h) and 4-8 h postdose], 2 (predose, 2-4 h and 6-8 h postdose), and 3 (predose and 2-8 h postdose) of Day 1 of each 28-day cycle
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable data for Cav,ss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/liter (nmol/L)
Arm/Group | Enzastaurin
Number analyzed (Participants) | 56
nanomoles/liter (nmol/L)
  Enzastaurin | 627 (74.4)
  Total analytes | 1160 (58.4)

ADVERSE EVENTS:
Time Frame: From randomization through 21 cycles (28-day cycle) and 30-day follow-up
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 20/60
Other Adverse Events (participants affected / at risk) | 54/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=60)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin (N=60)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Ascites (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 10 (11)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 8 (14)
Asthenia (General disorders) | 3 (3)
Fatigue (General disorders) | 9 (9)
Oedema peripheral (General disorders) | 4 (5)
Pyrexia (General disorders) | 7 (7)
Bronchitis (Infections and infestations) | 3 (3)
Haemoglobin (Investigations) | 3 (4)
Weight decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Chromaturia (Renal and urinary disorders) | 3 (3)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1/18 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (7)
Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days